CLINICAL TRIAL: NCT01644344
Title: Pilot Study for a Randomized Control Trial Comparing the Cost of a Simplified Post-Operative Radiographic (SPOR) Protocol for Fractures With Stable Internal Fixation Treated at Health Sciences Centre
Brief Title: A Prospective Trial Comparing the Cost of Post Operative X-rays for Fractures Treated With Stable Internal Fixation
Acronym: SPOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre Foundation, Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RI1211:135
Record Dates: First submitted 2012-07-12; First posted 2012-07-19 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-03

CONDITIONS: Simplified Postoperative Radiographs
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Who Masked: Care Provider

ARMS (2):
- X-ray (Active Comparator): Control group: patients will receive standard radiographs post-operative day one or two in hospital, as well as radiographs in clinic at two and six weeks. Each time radiographs are completed, the surgeon or resident will document if a change in fixation position is noted and if a change in patient management will be entertained (addition, modification or maintenance of cast or splint use, modification of or decision not to advance activity level, need for further surgery to adjust fixation or fracture reduction). The patients' time spent in clinic will be recorded upon arrival and upon completion of the patient-physician interaction.
  Interventions: Other: Xray
- No X-ray (Active Comparator)
  Interventions: Other: No-Xray

INTERVENTIONS:
Other: No-Xray — Treatment group: these patients will not have routine post-operative in hospital radiographs, or radiographs in clinic at two weeks. After examining the patient, the surgeon or resident can order radiographs if required at any time. The decision will be made based on patient complaints of increased pain, appearance of abuse of the splint or cast suggesting lack of compliance or visible clinical deformity of the limb. The reason leading to radiographs will be documented by the ordering physician. If radiographs are ordered based on a wound complication, this will be specifically documented. Radiographic findings will be documented on a form identical to that used for the control group.
  Arms: No X-ray
Other: Xray
  Arms: X-ray

SUMMARY:
The standard post-operative radiographic protocol for the monitoring of fractures at HSC includes post-operative in hospital radiographs as well as radiographs at the two week follow up appointment. This is in addition to good quality intra-operative radiographs. With current operative techniques and implants, orthopaedic surgeons can achieve reliably stable internal fixation. In fact, patients are often allowed to take weight through the fractured limb immediately post-operatively. In these cases, redundant post-operative radiographs likely represent an avoidable cost to the system financially, and an avoidable cost to the patient in additional time spent in hospital and unnecessary radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

* Femur fracture treated with intramedullary nailing
* Tibia fracture treated with intramedullary nailing
* Ankle fractures treated with standard compression technique
* Humeral shaft fractures treated with standard compression technique
* Forearm fractures treated with standard compression technique
* One or both bones fractured
* Simple fracture or presence of single butterfly fragment treated with lag screw
* Clavicle fracture treated with standard compression technique
* Olecranon fracture treated with standard compression technique

Exclusion Criteria:

* Age < 17 years, or open growth plates
* Multiple orthopaedic fractures
* History of radiographic appearance of osteoporosis or osteopenia or poor operative bone quality
* Likely difficult with follow-up in first 6 weeks
* Same day surgery case
* Surgeon feels patient should be excluded

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
cost-effectiveness of a simplified post-operative radiographic protocol for selected fractures | post-operative day one or two in hospital, as well as in clinic at two and six weeks
  Cost-effectiveness will be measured by calculating cost of x-ray, patient care and time spent by patient in clinic.

SECONDARY OUTCOMES:
Patient satisfaction | At six weeks post-op
  Validated Patient Satisfaction Questionnaire to be used to measure patient satisfaction with a simplified post-operative radiographic protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada